CLINICAL TRIAL: NCT01454817
Title: A Study of Symptoms and Quality of Life in Patients With ICDs and Their Caregivers
Brief Title: A Study of Symptoms and Quality of Life in Patients With Implantable Cardiac Defibrillators (ICDs) and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HSM 10-00041
Record Dates: First submitted 2011-10-14; First posted 2011-10-19 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Quality of Life; Implantable Cardiac Defibrillators; ICDs
Keywords: Quality of Life; Implantable Cardiac Defibrillators; ICDs
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with ICDs (Other)
  Interventions: Behavioral: Quality of life
- Caregivers of Patients with ICDs (Other)
  Interventions: Behavioral: Quality of life

INTERVENTIONS:
Behavioral: Quality of life — Improving Quality of Life

SUMMARY:
The purpose of this study is to better understand symptoms and quality of life in patients with heart disease and implantable defibrillators (ICDs).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patient has an ICD
* Age > 18
* Fluent in English
* Consistent and reliable access to a phone.

Caregivers of Patients:

* Age > 18
* Fluent in English
* Consistent and reliable access to a phone

Exclusion Criteria:

* Not having an ICD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Actual)
Dates: Start 2012-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Physical Symptoms | every 3 months plus after hospitalizations for an average of 1 year
  physical symptoms of pain, shortness of breath, depression, anxiety
Psychological Symptoms | every 3 months plus after hospitalizations for an average of 1 year
  Psychological symptoms of anxiety and depression

SECONDARY OUTCOMES:
Quality of Life | every 3 months plus after hospitalizations for an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Goldstein, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - University of Colorado - Denver, Denver, Colorado
  - Yale New-Haven Hospital, New Haven, Connecticut
  - Mayo Medical Center, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania